CLINICAL TRIAL: NCT06347432
Title: Em-power: Maximizing Functional Independence for Children With Severe Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Grand Valley State University (Other)
Responsible Party: Principal Investigator, Lisa Kenyon, Professor, Grand Valley State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-119-H
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Experimental Group (Experimental): Group A: The Experimental Group will receive the 8-week evidence-based PWC skills training using the IndieTrainer System following T0 baseline testing
  Interventions: Other: Power wheelchair skills training using the IndieTrainer system
- Group B: Wait List Control Group (No Intervention): Group B: The Wait List Control Group will receive the 8-week evidence-based PWC skills training using the IndieTrainer System following T2 testing

INTERVENTIONS:
Other: Power wheelchair skills training using the IndieTrainer system — The IndieTrainer system will be used to provide the power wheelchair (PWC) skills training sessions. The IndieTrainer is comprised of a mobility device and an array of video-based gamified training modules designed to facilitate PWC training. The IndieTrainer mobility device temporarily converts a manual wheelchair into a powered wheelchair, thereby allowing children to remain in their own manual wheelchair and use their own custom seating system during power wheelchair skills training activities. Principles outlined in the Assessment of Learning Powered mobility use (ALP) Facilitating Strategies for each ALP Assessment phase will guide the intervention sessions.
  Arms: Group A: Experimental Group

SUMMARY:
For children with severe cerebral palsy, a powered wheelchair (PWC) may provide their only option for functional mobility and independence. PWC use is often restricted to a small percentage of children who can quickly demonstrate proficient PWC skills within a single 30-minute PWC trial. This 2-arm, parallel group, single blinded, pre-test-post-test randomized controlled trial will test our hypothesis that an 8-week PWC skills training intervention will produce greater improvements in children's PWC skills capacity immediately after the intervention and at an 8-week follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe CP (Gross Motor Function Classification System Level IV or V)
* Inability to functionally walk or functionally propel a manual wheelchair as assessed by the Principal Investigator a licensed physical therapist
* Demonstrate cause and effect skills in the IndieTrainer consistent with an Assessment of Learning Powered mobility use (ALP Assessment) Phase 4 or higher (i.e., understand that they are moving the IndieTrainer using the switch(es) or joystick) as assessed by the Principal Investigator, a licensed physical therapist.
* In addition, one parent/caregiver must be conversant in English and be able to provide their child's medical and health history and be willing to take on the parent participant role.

Exclusion Criteria:

* The inability to sit in their own manual wheelchair or adaptive stroller for 60 minutes (as this would preclude them safely using the IndieTrainer System for the 60-minute intervention sessions)
* Their manual wheelchair or adaptive stroller cannot be safely used with the IndieTrainer System
* They already have an individually prescribed power wheelchair
* If the Principal Investigator, a licensed physical therapist, determines that based on the child's medical and health history, that they cannot safely participate in power wheelchair skills training.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in understanding how to use a power wheelchair | Baseline (T0) pre-intervention, immediately after the conclusion of the 8-week intervention period (T1), and at the single session retention trial 8 weeks after the end of the intervention period (T2)
  This outcome will be assessed using each participant's score (from a low of Phase 1 to a high of Phase 8) on the Assessment of Learning Powered mobility use. The Assessment of Learning Powered mobility use (ALP) is a process-based measure detailing 8 phases of learning (Phase 1 - Novice to Phase 8 - Expert) within 3 stages: Stage 1 - the Introvert Stage where the child focuses on exploring cause and effect within the function of the power mobility device; Stage 2 - the Explore Sequencing Stage where the child focuses on how to sequence the operations to maneuver the power mobility device; and Stage 3 - the Extrovert Stage where the child is focused on using the power mobility device in daily life. Higher scores therefore indicate a better outcome.
Change in power wheelchair skill performance | Baseline (T0) pre-intervention, immediately after the conclusion of the 8-week intervention period (T1), and at the single session retention trial 8 weeks after the end of the intervention period (T2)
  This outcome will be assessed using the Wheelchair Skills Checklist, a task-based measure that evaluates a child's performance of 7 specific power mobility skills using a 3-point ordinal scale from 0-2 where a score of "0" indicates the participant Does Not Perform the skill, a score of "1" indicates that the skill is Emerging, and a score of "2" indicates the participant Performs the Skill. Higher scores therefore indicate a better outcome.

SECONDARY OUTCOMES:
Change in parental/caregiver perceptions of changes in their children's performance of power wheelchair skill performance | Baseline (T0) pre-intervention and immediately after the conclusion of the 8-week intervention period (T1)
  This outcome will be assessed using the Canadian Occupational Performance Measure to identify, prioritize, and rate parent/caregiver perceptions of children's performance of power wheelchair skills. A total of 4-5 occupational performance issues in the area of power wheelchair skills will be identified and scored on a 1-10 scale, where a "1" is the lowest score and a "10 is the highest score, for both the caregiver's perception of the child's performance and their satisfaction with the child's performance.
Change in children's perceptions of changes in their performance of power wheelchair skill performance | Baseline (T0) pre-intervention and immediately after the conclusion of the 8-week intervention period (T1)
  This outcome will be assessed using the Canadian Occupational Performance Measure to identify, prioritize, and rate child perceptions of their performance of power wheelchair skills. A total of 4-5 occupational performance issues in the area of power wheelchair skills will be identified and scored on a 1-10 scale, where a "1" is the lowest score and a "10 is the highest score, for both the child's perception of their performance and their satisfaction with their performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Grand Valley State University, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
This study is being funded by the National Institutes of Health (NIH). The NIH requires that research data collected in this study be made available to other researchers. As such, the de-identified data collected in this study will be placed in a repository where it can be accessed by other researchers for future studies.